CLINICAL TRIAL: NCT01231412
Title: A Randomized Phase III Study to Determine the Most Promising Postgrafting Immunosuppression for Prevention of Acute GVHD After Unrelated Donor Hematopoietic Cell Transplantation Using Nonmyeloablative Conditioning for Patients With Hematologic Malignancies: A Multi-center Trial
Brief Title: Graft-Versus-Host Disease Prophylaxis in Treating Patients With Hematologic Malignancies Undergoing Unrelated Donor Peripheral Blood Stem Cell Transplant
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Brenda Sandmaier, Principal Investigator, Fred Hutchinson Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2448.00; NCI-2010-02035 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2448.00 (Other: Fred Hutch/University of Washington Cancer Consortium); P01CA018029 (NIH); P30CA015704 (NIH)
Record Dates: First submitted 2010-10-28; First posted 2010-11-01 (Estimated); Results first posted 2017-12-04 (Actual); Last update posted 2019-10-24 (Actual); Status verified 2019-10

CONDITIONS: Acute Lymphoblastic Leukemia; Acute Myeloid Leukemia; Aggressive Non-Hodgkin Lymphoma; Chronic Lymphocytic Leukemia; Diffuse Large B-Cell Lymphoma; Hematopoietic and Lymphoid Cell Neoplasm; Indolent Non-Hodgkin Lymphoma; Mantle Cell Lymphoma; Myelodysplastic Syndrome; Myeloproliferative Neoplasm; Prolymphocytic Leukemia; Recurrent Chronic Lymphocytic Leukemia; Recurrent Plasma Cell Myeloma; Refractory Chronic Lymphocytic Leukemia; Refractory Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Refractory Hodgkin Lymphoma; Small Lymphocytic Lymphoma; T-Cell Chronic Lymphocytic Leukemia; Waldenstrom Macroglobulinemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Large B-Cell, Diffuse; Hematologic Neoplasms; Lymphoma, Mantle-Cell; Myelodysplastic Syndromes; Myeloproliferative Disorders; Leukemia, Prolymphocytic; Multiple Myeloma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Hodgkin Disease; Leukemia, Prolymphocytic, T-Cell; Waldenstrom Macroglobulinemia | interventions — Cyclosporine; Cyclosporins; fludarabine phosphate; Mycophenolic Acid; Peripheral Blood Stem Cell Transplantation; Sirolimus; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm I (MMF and CSP) (Active Comparator): Patients receive FLU IV over 30 minutes on days -4 to -2. Patients also receive CSP PO BID on days -3 to 96 with taper to day 150 and MMF PO TID daily on days 0-29 and then BID on days 30-150 with taper to day 180. Patients undergo allogeneic PBSCT on day 0 following the TBI.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Cyclosporine; Drug: Fludarabine Phosphate; Drug: Mycophenolate Mofetil; Procedure: Peripheral Blood Stem Cell Transplantation; Radiation: Total-Body Irradiation
- Arm II (MMF, CSP, and Sirolimus) (Experimental): Patients receive FLU and CSP as in Arm I and sirolimus PO QD on days -3 to 150 with taper to day 180. Patients also receive MMF PO TID on days 0-29 and then BID on days 30-40. MMF will then be discontinued without taper unless GVHD or disease relapse/progression occurs. Patients undergo allogeneic PBSCT on day 0 following the TBI.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Cyclosporine; Drug: Fludarabine Phosphate; Drug: Mycophenolate Mofetil; Procedure: Peripheral Blood Stem Cell Transplantation; Drug: Sirolimus; Radiation: Total-Body Irradiation
- Arm 0 (CSP and Sirolimus) (Experimental): Patients receive CSP orally (PO) twice daily (BID) on days -3 to 96 with taper to day 150 and and sirolimus PO once daily (QD) on days -3 to 150 with taper to day 180. Arm removed as of 14-Sep-2011
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Cyclosporine; Drug: Fludarabine Phosphate; Procedure: Peripheral Blood Stem Cell Transplantation; Drug: Sirolimus; Radiation: Total-Body Irradiation

INTERVENTIONS:
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo allogeneic PBSCT
  Other Names: allogeneic stem cell transplantation; HSC; HSCT
Drug: Cyclosporine — Given PO or IV
  Other Names: 27-400; Ciclosporin; CsA; Cyclosporin; Cyclosporin A; Gengraf; Neoral; OL 27-400; Sandimmun; Sandimmune; SangCya
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; SH T 586
Drug: Mycophenolate Mofetil — Given PO
  Other Names: Cellcept; MMF
  Arms: Arm I (MMF and CSP); Arm II (MMF, CSP, and Sirolimus)
Procedure: Peripheral Blood Stem Cell Transplantation — Undergo allogeneic PBSCT
  Other Names: PBPC transplantation; Peripheral Blood Progenitor Cell Transplantation; Peripheral Stem Cell Support; Peripheral Stem Cell Transplantation
Drug: Sirolimus — Given PO
  Other Names: AY 22989; RAPA; Rapamune; RAPAMYCIN; SILA 9268A; WY-090217
  Arms: Arm 0 (CSP and Sirolimus); Arm II (MMF, CSP, and Sirolimus)
Radiation: Total-Body Irradiation — Undergo TBI
  Other Names: TOTAL BODY IRRADIATION; Whole-Body Irradiation

SUMMARY:
This randomized phase III trial studies how well graft-vs-host disease (GVHD) prophylaxis works in treating patients with hematologic malignancies undergoing unrelated donor peripheral blood stem cell transplant. Giving chemotherapy and total-body irradiation before a donor peripheral blood stem cell transplant (PBSCT) helps stop the growth of cancer cells. It may also stop the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Giving total-body irradiation (TBI) together with fludarabine phosphate (FLU), cyclosporine (CSP), mycophenolate mofetil (MMF), or sirolimus before transplant may stop this from happening.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the effectiveness of 2 GVHD prophylaxis regimens in preventing acute grades II-IV GVHD.

SECONDARY OBJECTIVES:

I. Compare non-relapse mortality in the 2 arms.

II. Compare survival and progression-free survivals in the 2 arms.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

All patients receive FLU intravenously (IV) over 30 minutes on days -4 to -2 followed by 2-3 Gy TBI on day 0.

ARM 0: Patients receive CSP orally (PO) twice daily (BID) on days -3 to 96 with taper to day 150 and and sirolimus PO once daily (QD) on days -3 to 150 with taper to day 180. Arm removed as of 14-Sep-2011

ARM I: Patients receive CSP orally (PO) twice daily (BID) on days -3 to 96 with taper to day 150 and MMF PO three times daily (TID) on days 0-29 and then BID on days 30-150 with taper to day 180.

ARM II: Patients receive CSP as in Arm I and sirolimus PO once daily (QD) on days -3 to 150 with taper to day 180. Patients also receive MMF PO TID on days 0-29 and then BID on days 30-40. MMF will then be discontinued without taper unless GVHD or disease relapse/progression occurs.

TRANSPLANTATION: Patients undergo allogeneic PBSCT on day 0 following the TBI.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Ages > 50 years with hematologic malignancies treatable by unrelated hematopoietic cell transplant (HCT)
* Ages =< 50 years of age with hematologic diseases treatable by allogeneic HCT who through pre-existing medical conditions or prior therapy are considered to be at high risk for regimen related toxicity associated with a high dose transplant (> 40% risk of transplant related mortality [TRM]); this criterion can include patients with a HCT-comorbidity index (CI) score of >= 1; transplants should be approved for these inclusion criteria by the principal investigators at the collaborating centers and at the Fred Hutchinson Cancer Research Center (FHCRC); all children < 12 years must be discussed with the FHCRC principal investigator (PI) prior to registration
* Ages =< 50 years of age with chronic lymphocytic leukemia (CLL)
* Ages =< 50 years of age with hematologic diseases treatable by allogeneic HCT who refuse a high-dose HCT; transplants must be approved for these inclusion criteria by the principal investigators at the collaborating centers and at FHCRC
* The following diseases will be permitted although other diagnoses can be considered if approved by Patient Care Conference (PCC) or the participating institutions' patient review committees and the principal investigators

  * Aggressive non-Hodgkin lymphomas (NHL) and other histologies such as diffuse large B cell NHL: not eligible for autologous HCT, not eligible for high-dose allogeneic HCT, or after failed autologous HCT
  * Mantle cell NHL: may be treated in first complete remission (CR); (diagnostic lumbar puncture [LP] required pre-transplant)
  * Low grade NHL: with < 6 month duration of CR between courses of conventional therapy
  * CLL: must have either:

    * Failed to meet National Cancer Institute (NCI) Working Group criteria for complete or partial response after therapy with a regimen containing FLU (or another nucleoside analog, e.g. 2-Chlorodeoxyadenosine [2-CDA], pentostatin) or experience disease relapse within 12 months after completing therapy with a regimen containing FLU (or another nucleoside analog);
    * Failed FLU-cyclophosphamide (CY)-Rituximab (FCR) combination chemotherapy at any time point; or
    * Have "17p deletion" cytogenetic abnormality; patients should have received induction chemotherapy but could be transplanted in 1st CR; or
    * Patients with a diagnosis of CLL (or small lymphocytic lymphoma) or diagnosis of CLL that progresses to prolymphocytic leukemia (PLL), or T-cell CLL or PLL
  * Hodgkin lymphoma: must have received and failed frontline therapy
  * Multiple myeloma: must have received prior chemotherapy; consolidation of chemotherapy by autografting prior to nonmyeloablative HCT is permitted
  * Acute myeloid leukemia (AML): must have < 5% marrow blasts at the time of transplant
  * Acute lymphocytic leukemia (ALL): must have < 5% marrow blasts at the time of transplant
  * Chronic myeloid leukemia (CML): patients in 1st chronic phase (CP1) must have failed or be intolerant of tyrosine-kinase inhibitors (TKI); patients beyond CP1 will be accepted if they have < 5% marrow blasts at time of transplant
  * Myelodysplasia (MDS)/myeloproliferative syndrome (MPS): patients must have < 5% marrow blasts at time of transplant
  * Waldenstrom's macroglobulinemia: must have failed 2 courses of therapy
* DONOR: FHCRC matching allowed will be grades 1.0 to 2.1: Unrelated donors who are prospectively:

  * Matched for human leukocyte antigen (HLA)-A, B, C, DRB1 and DQB1 by high resolution typing
  * Only a single allele disparity will be allowed for HLA-A, B, or C as defined by high resolution typing
* DONOR: Donors are excluded when preexisting immunoreactivity is identified that would jeopardize donor hematopoietic cell engraftment; this determination is based on the standard practice of the individual institution; the recommended procedure for patients with 10 of 10 HLA allele level (phenotypic) match is to obtain a panel reactive antibody (PRA) screens to class I and class II antigens for all patients before HCT; if the PRA shows > 10% activity, then flow cytometric or B and T cell cytotoxic cross matches should be obtained; the donor should be excluded if any of the cytotoxic cross match assays are positive; for those patients with an HLA class I allele mismatch, flow cytometric or B and T cell cytotoxic cross matches should be obtained regardless of the PRA results; a positive anti-donor cytotoxic crossmatch is an absolute donor exclusion
* DONOR: Patient and donor pairs homozygous at a mismatched allele in the graft rejection vector are considered a two-allele mismatch, i.e., the patient is A*0101 and the donor is A*0102, and this type of mismatch is not allowed
* DONOR: Only filgrastim (G-CSF) mobilized PBSC only will be permitted as a hematopoietic stem cell (HSC) source on this protocol

Exclusion Criteria:

* Patients with rapidly progressive intermediate or high grade NHL
* Patients with a diagnosis of chronic myelomonocytic leukemia (CMML)
* Patients with refractory anemia with excess blasts (RAEB) who have not received myelosuppressive chemotherapy i.e. induction chemotherapy
* Central nervous system (CNS) involvement with disease refractory to intrathecal chemotherapy
* Presence of circulating leukemic blasts (in the peripheral blood) detected by standard pathology for patients with AML, ALL or CML
* Presence of >= 5% circulating leukemic blasts (in the peripheral blood) detected by standard pathology for patients with MDS/MPS
* Fertile men or women unwilling to use contraceptive techniques during and for 12 months following treatment
* Females who are pregnant or breast-feeding
* Patients with active non-hematological malignancies (except non-melanoma skin cancers) or those with non-hematological malignancies (except non-melanoma skin cancers) who have been rendered with no evidence of disease, but have a greater than 20% chance of having disease recurrence within 5 years; this exclusion does not apply to patients with non-hematologic malignancies that do not require therapy
* Fungal infections with radiological progression after receipt of amphotericin B or active triazole for greater than 1 month
* Cardiac ejection fraction < 35% (or, if unable to obtain ejection fraction, shortening fraction of < 26%); ejection fraction is required if age > 50 years or there is a history of anthracycline exposure or history of cardiac disease; patients with a shortening fraction < 26% may be enrolled if approved by a cardiologist
* Diffusing capacity of the lung for carbon monoxide (DLCO) < 40%, total lung capacity (TLC) < 40%, forced expiratory volume in one second (FEV1) < 40% and/or receiving supplementary continuous oxygen
* The FHCRC PI of the study must approve of enrollment of all patients with pulmonary nodules
* Patients with clinical or laboratory evidence of liver disease would be evaluated for the cause of liver disease, its clinical severity in terms of liver function, and the degree of portal hypertension; patients will be excluded if they are found to have fulminant liver failure, cirrhosis of the liver with evidence of portal hypertension, alcoholic hepatitis, esophageal varices, a history of bleeding esophageal varices, hepatic encephalopathy, uncorrectable hepatic synthetic dysfunction evinced by prolongation of the prothrombin time, ascites related to portal hypertension, bridging fibrosis, bacterial or fungal liver abscess, biliary obstruction, chronic viral hepatitis with total serum bilirubin > 3 mg/dL, or symptomatic biliary disease
* Karnofsky scores < 60 or Lansky Score < 50
* Patient has poorly controlled hypertension and on multiple antihypertensives
* Human immunodeficiency virus (HIV) positive patients
* Active bacterial or fungal infections unresponsive to medical therapy
* All patients receiving antifungal therapy voriconazole, posaconazole, or fluconazole and who are then randomized to ARM 2 must have sirolimus reduced according to the Standard Practice Antifungal Therapy Guidelines
* The addition of cytotoxic agents for "cytoreduction" with the exception of tyrosine kinase inhibitors (such as imatinib), cytokine therapy, hydroxyurea, low dose cytarabine, chlorambucil, or Rituxan will not be allowed within three weeks of the initiation of conditioning
* DONOR: Donor (or centers) who will exclusively donate marrow
* DONOR: Donors who are HIV-positive and/or, medical conditions that would result in increased risk for G-CSF mobilization and harvest of PBSC

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2010-11; Primary Completion 2016-10-08 (Actual); Study Completion 2017-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brenda Sandmaier, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (11):
- United States (6):
  - University of Colorado, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Emory University/Winship Cancer Institute, Atlanta, Georgia
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - VA Puget Sound Health Care System, Seattle, Washington
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington
- Denmark (2):
  - Aarhus University Hospital, Aarhus
  - Rigshospitalet University Hospital, Copenhagen
- Germany (3):
  - Medizinische Univ Klinik Koln, Cologne
  - Universitaet Leipzig, Leipzig
  - University of Tuebingen-Germany, Tübingen

REFERENCES:
- [Derived] Cooper JP, Storer BE, Granot N, Gyurkocza B, Sorror ML, Chauncey TR, Shizuru J, Franke GN, Maris MB, Boyer M, Bruno B, Sahebi F, Langston AA, Hari P, Agura ED, Lykke Petersen S, Maziarz RT, Bethge W, Asch J, Gutman JA, Olesen G, Yeager AM, Hubel K, Hogan WJ, Maloney DG, Mielcarek M, Martin PJ, Flowers MED, Georges GE, Woolfrey AE, Deeg JH, Scott BL, McDonald GB, Storb R, Sandmaier BM. Allogeneic hematopoietic cell transplantation with non-myeloablative conditioning for patients with hematologic malignancies: Improved outcomes over two decades. Haematologica. 2021 Jun 1;106(6):1599-1607. doi: 10.3324/haematol.2020.248187. PMID 32499241
- [Derived] Sandmaier BM, Kornblit B, Storer BE, Olesen G, Maris MB, Langston AA, Gutman JA, Petersen SL, Chauncey TR, Bethge WA, Pulsipher MA, Woolfrey AE, Mielcarek M, Martin PJ, Appelbaum FR, Flowers MED, Maloney DG, Storb R. Addition of sirolimus to standard cyclosporine plus mycophenolate mofetil-based graft-versus-host disease prophylaxis for patients after unrelated non-myeloablative haemopoietic stem cell transplantation: a multicentre, randomised, phase 3 trial. Lancet Haematol. 2019 Aug;6(8):e409-e418. doi: 10.1016/S2352-3026(19)30088-2. Epub 2019 Jun 24. PMID 31248843

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (MMF and CSP) | Arm II (MMF, CSP, and Sirolimus) | Arm 0 (CSP and Sirolimus)
Started | 77 | 91 | 6
Completed | 77 | 90 | 6
Not Completed | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (MMF and CSP) | Arm II (MMF, CSP, and Sirolimus) | Arm 0 (CSP and Sirolimus) | Total
Number analyzed (Participants) | 77 | 91 | 6 | 174
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 52 | 50 | 4 | 106
  >=65 years | 25 | 41 | 2 | 68
Age, Continuous [Median (Full Range); unit: years] | 61.94 [18.2 to 77.09] | 63.75 [41.02 to 79] | 59.515 [36.47 to 67.83] | 62.655 [18.2 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 28 | 2 | 57
  Male | 50 | 63 | 4 | 117
Region of Enrollment [Number; unit: participants]
  United States | 65 | 78 | 6 | 149
  Denmark | 10 | 12 | 0 | 22
  Germany | 2 | 1 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Grades II-IV Acute GVHD
Description: Number of patients with grades II-IV acute GVHD
  aGVHD Stages
  Skin:
  1. a maculopapular eruption involving < 25% BSA
  2. a maculopapular eruption involving 25 - 50% BSA
  3. generalized erythroderma
  4. generalized erythroderma w/ bullous formation and often w/ desquamation
  Liver:
  1. bilirubin 2.0 - 3.0 mg/100 mL
  2. bilirubin 3 - 5.9 mg/100 mL
  3. bilirubin 6 - 14.9 mg/100 mL
  4. bilirubin > 15 mg/100 mL
  Gut:
  Diarrhea is graded 1 - 4 in severity. Nausea and vomiting and/or anorexia caused by GVHD is assigned as 1 in severity. The severity of gut involvement is assigned to the most severe involvement noted. Patients w/ visible bloody diarrhea are at least stage 2 gut and grade 3 overall.
  aGVHD Grades Grade II: Stage 1 - 2 skin w/ no gut/liver involvement Grade III: Stage 2 - 4 gut involvement and/or stage 2 - 4 liver involvement Grade IV: Pattern and severity of GVHD similar to grade 3 w/ extreme constitutional symptoms or death
Time Frame: At day 100 post-transplant
Population: One subject on Arm II aborted transplant during conditioning and subsequently went on to transplant on a different study. This subject was counted towards accrual but not evaluated with respect to outcome measures.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (MMF and CSP) | Arm II (MMF, CSP, and Sirolimus) | Arm 0 (CSP and Sirolimus)
Number analyzed (Participants) | 77 | 90 | 6
Participants | 39 | 22 | 3

2. Secondary Outcome: Number of Patients With Chronic Extensive GVHD
Description: Number of patients who developed chronic extensive GVHD post-transplant. The diagnosis of chronic GVHD requires at least one manifestation that is distinctive for chronic GVHD as opposed to acute GVHD. In all cases, infection and others causes must be ruled out in the differential diagnosis of chronic GVHD.
Time Frame: Up to 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (MMF and CSP) | Arm II (MMF, CSP, and Sirolimus) | Arm 0 (CSP and Sirolimus)
Number analyzed (Participants) | 77 | 90 | 6
Participants | 38 | 43 | 3

3. Secondary Outcome: Number of Patients With Grades III-IV Acute GVHD
Description: Number of patients with grades III-IV acute GVHD
  aGVHD Stages
  Skin:
  1. a maculopapular eruption involving < 25% BSA
  2. a maculopapular eruption involving 25 - 50% BSA
  3. generalized erythroderma
  4. generalized erythroderma w/ bullous formation and often w/ desquamation
  Liver:
  1. bilirubin 2.0 - 3.0 mg/100 mL
  2. bilirubin 3 - 5.9 mg/100 mL
  3. bilirubin 6 - 14.9 mg/100 mL
  4. bilirubin > 15 mg/100 mL
  Gut:
  Diarrhea is graded 1 - 4 in severity. Nausea and vomiting and/or anorexia caused by GVHD is assigned as 1 in severity. The severity of gut involvement is assigned to the most severe involvement noted. Patients w/ visible bloody diarrhea are at least stage 2 gut and grade 3 overall.
  aGVHD Grades Grade II: Stage 1 - 2 skin w/ no gut/liver involvement Grade III: Stage 2 - 4 gut involvement and/or stage 2 - 4 liver involvement Grade IV: Pattern and severity of GVHD similar to grade 3 w/ extreme constitutional symptoms or death
Time Frame: Up to 100 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (MMF and CSP) | Arm II (MMF, CSP, and Sirolimus) | Arm 0 (CSP and Sirolimus)
Number analyzed (Participants) | 77 | 90 | 6
Participants | 8 | 2 | 0

4. Secondary Outcome: Number of Non-Relapse Mortalities
Description: Number of subjects expired without disease progression/relapse.
Time Frame: Up to 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (MMF and CSP) | Arm II (MMF, CSP, and Sirolimus) | Arm 0 (CSP and Sirolimus)
Number analyzed (Participants) | 77 | 90 | 6
Participants | 12 | 4 | 0

5. Secondary Outcome: Number of of Participants Surviving Overall
Description: Number of subjects surviving overall post-transplant.
Time Frame: Up to 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (MMF and CSP) | Arm II (MMF, CSP, and Sirolimus) | Arm 0 (CSP and Sirolimus)
Number analyzed (Participants) | 77 | 90 | 6
Participants | 53 | 75 | 6

6. Secondary Outcome: Number of Participants With Relapse/Progression
Description: Relapse/Progression criteria:
  CML New cytogenetic abnormality and/or development of accelerated phase or blast crisis. The criteria for accelerated phase will be defined as unexplained fever >38.3°C, new clonal cytogenetic abnormalities in addition to a single Ph-positive chromosome, marrow blasts and promyelocytes >20%.
  AML, ALL, MDS >5% blasts by morphologic or flow cytometric evaluation of the BMA or appearance of extramedullary disease CLL ≥1 of: Physical exam/imaging studies ≥50% increase or new, circulating lymphocytes by morphology and/or flow cytometry ≥50% increase, and lymph node biopsy w/ Richter's transformation.
  NHL >25% increase in the sum of the products of the perpendicular diameters of marker lesions, or the appearance of new lesions.
  MM
  ≥100% increase of the serum myeloma protein from its lowest level, or reappearance of myeloma peaks that had disappeared w/ treatment; or definite increase in the size or numb
Time Frame: Up to 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (MMF and CSP) | Arm II (MMF, CSP, and Sirolimus) | Arm 0 (CSP and Sirolimus)
Number analyzed (Participants) | 77 | 90 | 6
Participants | 16 | 16 | 1

ADVERSE EVENTS:
Time Frame: AEs: Conditioning through Day 100; SAEs: Conditioning through Day 200
Arm/Group | Arm I (MMF and CSP) | Arm II (MMF, CSP, and Sirolimus) | Arm 0 (CSP and Sirolimus)
Serious Adverse Events (participants affected / at risk) | 0/77 | 0/90 | 0/6
Other Adverse Events (participants affected / at risk) | 27/77 | 26/90 | 3/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (MMF and CSP) (N=77) | Arm II (MMF, CSP, and Sirolimus) (N=90) | Arm 0 (CSP and Sirolimus) (N=6)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 3 (3) | 0 (0)
"Adult respiratory distress syndrome" (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Allergic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 7 (7) | 1 (1) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Colonic hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 4 (4) | 4 (4) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Encephalitis infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 6 (7) | 3 (3) | 0 (0)
Fecal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hemolysis (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 4 (4) | 0 (0)
Hypotension (Vascular disorders) | 2 (3) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (4) | 0 (0)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Renal and urinary disorders - Other (Hemorrhagic cystitis) (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Thromboembolic event (Vascular disorders) | 2 (3) | 1 (2) | 0 (0)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Weight loss (Investigations) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-20): https://cdn.clinicaltrials.gov/large-docs/12/NCT01231412/Prot_SAP_000.pdf